CLINICAL TRIAL: NCT06745245
Title: Effect of Oral Consumption of a Symbiotic Gelatin on the Presence of Gastrointestinal Symptoms and Quality of Life in People With Chronic Kidney Disease Grades G3a, G3b, G4, G5 and G5D in Mexico
Brief Title: Effect of Oral Consumption of a Symbiotic Gelatin on the Presence of Gastrointestinal Symptoms and Quality of Life in People With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NIN Institute (Industry)
Collaborators: Centro Medico Issemym (Other)
Responsible Party: Principal Investigator, Ari Cisneros-Hernández, Principal Investigator, NIN Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI0003/24
Record Dates: First submitted 2024-10-18; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Disease(CKD); Dysbiosis Symptoms Linked to Pathology; Probiotics Supplement
Keywords: chronic kidney disease; probiotics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Nutrition Assessment; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: In the intervention, the specialized oral supplement plus very general nutritional advice is provided, to the participants in the different stages of kidney disease, as well as in the presence of replacement therapy, laboratory studies (blood and urine) are indicated to all groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Arm Intervention (Experimental): Intervention group: The specialized oral supplement is provided, with the consumption of 1 dose (15 g) per day along with individualized nutritional advice. For 1.5 months
  Interventions: Dietary Supplement: Nutritional counseling and supplementation with a gelatin with prebiotic fiber and probiotic microorganisms

INTERVENTIONS:
Dietary Supplement: Nutritional counseling and supplementation with a gelatin with prebiotic fiber and probiotic microorganisms — One serving (15 g) of symbiotic gelatin
  Other Names: Symbiotic gelatin

SUMMARY:
In patients with chronic kidney disease (CKD) there is a high prevalence of gastrointestinal disorders and negative changes in the microbiota and assimilation of nutrients, which is associated with an increased risk of morbidity and mortality.

DETAILED DESCRIPTION:
Gastrointestinal changes in CKD. In addition to the intrinsic effect of CKD on the gastrointestinal tract, extrinsic factors such as;Changes in diet (reduction in fiber consumption and increase in ultra-processed products), decrease in physical activity which impacts the reduction of gastrointestinal motility and the consumption of medications constantly can affect the structure and function at the gastrointestinal level. In HD patients without diabetes mellitus, the prevalence of dyspepsia is 40% to 70%. It is hypothesized that the pathophysiology of functional dyspepsia is multifactorial and may include a number of factors such as; abnormal gastric motility, impaired visceral sensation, dysregulation of the gut-brain axis, and low-grade inflammation.

Clinical evidence supports the theory that gut with dysbiosis contributes significantly to the deterioration of CKD progression, leading to an increase in bowel-derived uremic toxins (GDUT) and worsening of the same disease. Strategies based on interventions in the gut microbiota could contribute as preventive and therapeutic approaches to modulate the microbiota and its metabolites and thereby slow down the progression of CKD.

The origin of uremic toxins in CKD is multiple. The importance of the toxin generated by intestinal microbial metabolism is becoming more and more known. About 10 g of protein reaches the colon daily, where gut bacteria break it down into metabolites such as ammonium, amines, thiols, phenols, and indoles. These products of fermentation in the colon are eliminated in the feces, although some are absorbed and eliminated by the kidney, so they accumulate in CKD.

On the other hand, patients with CKD are constantly polymedicated. Some drugs frequently prescribed to these patients can alter the gut microbiota, especially antibiotics. There are also others that can slow down intestinal transit, phosphorus binders, ion exchange resins, or iron supplements, whose impact on the microbiota is not yet well known.

This project will provide practical information for the validation of the therapeutic effect of a symbiotic gelatin on gastrointestinal symptoms and quality of life in patients with CKD with and without replacement therapy, which will be useful both for health professionals and for the patients themselves.

MAIN OBJETIVE:

To evaluate the effect of oral consumption of synbiotic for one and a half months on the presence of gastrointestinal symptoms and the level of quality of life in people with CKD.

STUDIO DESING:

Controlled clinical trial with an intervention period of 1.5 months.

PROCESS:

1. Identify those patients who are candidates to participate in the clinical trial.
2. Review the inclusion and exclusion criteria.
3. Invite identified patients to participate in the clinical trial.

Full Assessment Nutritional Appointment - Nutritionist (Initial Consultation) Blood and urine sampling (if applicable and the patient still maintains diuresis), data capture, VGS, quality of life survey, the presence of general and gastrointestinal symptoms is evaluated, the Bristol scale is applied as well as anthropometric measurements. The first treatment is given with 15 sachets of the probiotic gel and indications are given for its consumption and storage.

(Monitoring week 1) A weekly telephone call to evaluate compliance with daily intakes, as well as to report the presence of gastrointestinal symptoms, findings of consumption, a product satisfaction scale is applied and the first educational material is sent (explanations are made and doubts are resolved). An appointment is scheduled for the next product delivery.

(Follow-up consultation) Delivery of the second box of treatment with 15 sachets again and the presence of gastrointestinal symptoms, findings on consumption and product satisfaction scale is reported.

(Monitoring week 3) A weekly telephone call to evaluate compliance with the daily intakes, as well as to report the presence of gastrointestinal symptoms, findings of consumption, a product satisfaction scale is applied and the second educational material is sent (explanations are made and doubts are resolved). An appointment is scheduled for the next product delivery.

(Follow-up consultation) Delivery of the third and last box of treatment with 15 sachets again and report the presence of gastrointestinal symptoms, findings to consumption and apply a product satisfaction scale.

(Monitoring week 5) A weekly telephone call to evaluate compliance with daily intakes, as well as to report the presence of gastrointestinal symptoms, findings of consumption, a product satisfaction scale is applied and the third educational material is sent (explanations are made and doubts are resolved) and an appointment is scheduled in the laboratory.

(Final consultation) Second and last appointment with the laboratory to take a blood and urine sample (if applicable and the patient still maintains diuresis), perform the capture of the final data, VGS, quality of life survey, evaluate the presence of general and gastrointestinal symptoms, apply the Bristol scale and take anthropometric measurements.

SAMPLE SIZE: 32 participants.

STATISTIC ANALYSIS:

The quantitative variables will be shown as mean and standard deviation or median and percentiles 25-75% depending on whether their distribution is normal or non-normal, and the qualitative variables will be represented in frequency and percentage. To test the normality of the variables, Shapiro Wilk tests will be performed. For the comparison of proportions between the groups, chi2 or Fisher's exact test will be carried out and to compare quantitative variables, Student's T or Mann-Whitney U will be used. For intragroup comparisons, Mc Nemar will be used for qualitative variables and ANOVA for repeated samples or Friedman's ANOVA for quantitative variables.

ELIGIBILITY:
Inclusion Criteria:

* Previous hospitalizations in the last month.
* Diagnosis of comorbidities such as cancer, decompensated heart failure, decompensated lung disease, decompensated liver disease, HIV, infection present within the last 3 months (chronic and/or acute) stroke, malabsorption syndrome or allergy to any ingredient of the nutritional supplement.
* Colon surgeries in the past 6 months (obstruction, resection of a portion).
* Presence of ostomies.
* Who show current treatment of antibiotics or oral iron.

Exclusion Criteria:

* Failure to attend evaluation and biochemical tests at the beginning and end of the study.
* Non-compliance with ≥ 10% of probiotics + fiber intakes (≥ 3 sachets in 15 days) during the intervention period.
* Identification of serious adverse effects.
* Withdrawal of voluntary participation by the patient.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | baseline intervention and 1.5 months
  Evaluate the presence and intesity of gastrointestinal symptoms for all patients from baseline to 1.5 month of intervention, through a Likert escale, with 5 being very intense and 1 being almost null.
Renal function | Baseline intervention and one and a half months
  Evaluate Glomerular Filtration Rate using the CKD-EPI creatinine equation in all patients at baseline and one and a half months

SECONDARY OUTCOMES:
Adherence to oral supplement | At 1.5 months of intervention
  Evaluate the level of adherence of all patients through a Likert scale, where 5 is very high adherence and 1 is very low adherence.
Adverse effects | At baseline and 1.5 months of intervention
  Evaluate the present and intensity of adverse effects during the intervention, through symptom assessment scale (SAS), where where 5 is very high intensity and 1 is very low

CONTACTS AND LOCATIONS:
Overall Officials: Paola Azucena Alvarado Pelayo, Bachelor, Principal Investigator — NIN Institute
Locations (1):
- Centro Médico Issemym, Toluca, Mexico

IPD SHARING:
Plan to Share IPD: No